CLINICAL TRIAL: NCT00610051
Title: Phase 3 Study of Alprostadil Continuous Intravenous Infusion to Maintain Clinical Stability in Severe Heart Failure Patients
Brief Title: ALP-1 Continuous Intravenous Infusion to Maintain Clinical Stability in Advanced Heart Failure
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Biopeutics Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3-T02-07-0106
Record Dates: First submitted 2008-01-14; First posted 2008-02-07 (Estimated); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: End Stage Cardiac Failure; HFrEF - Heart Failure With Reduced Ejection Fraction; NYHF Class III-IV
Keywords: advanced HFrEF
MeSH Terms: interventions — Alprostadil

STUDY DESIGN:
Intervention Model Description: This multicenter, double-blind, placebo-controlled, randomized, parallel-group trial will study up to approximately 400 patients with advanced HFrEF who are not expected to receive heart transplant or LVAD placement for 6 months after enrollment. Eligible patients will be randomized (1:1) to receive either alprostadil 250 μg/day, regardless of body weight, or placebo (normal saline) given in a continuous infusion. Primary objective is to evaluate the effect of continue alprostadil infsuion, 250 mcg/day on major outcome up to 6 months after randomization.
  Secondary Objectives are to assess the safety of continunous infsuion alprostadil 250mcg/day.
  Other Obectives are to evaluate the effictiveness and safety of continuous alprostadil infusion on other efficacy and patient health care related outcomes.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The party or parties involved in the study trials who are prevented from having knowledge of the interventions assigned to individual participants
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- trial arm (Active Comparator): 6 months central continuous infusion with Alp_1 by infusion pump.
  Interventions: Drug: Alprostadil
- Placebo arm (Placebo Comparator): 6 months central infusion with NS by infusion pump with exact infusion rat as trial arm.
  Interventions: Drug: Alprostadil

INTERVENTIONS:
Drug: Alprostadil — central venous access continuous delivery with 500mcg/48 hours in active arm

SUMMARY:
This is a global multicenter, doubleblind, placebo-controlled, randomized, parallel-group study that compares ALP-1 given in a continuous infusion ( compared to placebo), 250mcg/day on majore outcomes up to 6 months after randomization in participants with advanced HF with reduced ejection fraction(HFrEF).

DETAILED DESCRIPTION:
We anticipate needing to screen ca. 600 patients in order to ransomize our target sample size of 400 participants. Participants will be randomozed 1:1to receive either alprostadil or placebo. Based on prior data, we expect the 6-month event rate to be 64% in the control group and 47% in the intervention group.

The planned duration of following-up for each patient is 6 months on the randomized trial intervention and a final follow-up visit will be performed 30 days after stopping the trial intervention. Eligible patients will be randomzied via a centralized IXRS to eith alprstadil or placebo. The planned study dusration is approximately 3-4 years from first randomized patient to last patient.

When a participant is deemed eligible to participate in the trial, a central line which will be used for infusion of double-blind treatment will be inserted, if not already in place. Continue infusion delivery system will be operated by a pump.

Infusion of trial intervention will be initiated while the participant is in the hospital of infusion centre and the participant is to remain under observation for at least 8 hours for monitoring of vital signs and adverse event(AEs).

ELIGIBILITY:
1. Patients older than 18 years of age, of any gender/sex and race/ethnicity
2. Patients with a diagnosis of advanced HFrEF as evidenced by (all must apply):

   1. most recent LVEF( by conventional imaging method<30% which was mwasured within 3 months prior randomization.
   2. Nt-proBNP >1500 ng/L or BNP >300 ng/L at prior randomization
   3. New York Heart Association (NYHA) functional class IIIb or IV, i.e., chronic dyspnoea or fatigue at rest or with minimal exertion for at least one month prior to consent.
   4. Renal dysfunction reflected by a glomerular filtration rate (GFR) <60 mL/min approximated by the Modification of Diet in Renal Disease formula.
   5. A total symptom score of KCCQ of <70measure within 24 hours of randomization
   6. Patients on all appropriate recommended HF therapy.
3. Patient should not be receiving continuous or planned intermittent intravenous infusions with a positive inotropic or vasodilator drug in a non-hospitalized setting
4. Patients should not be considered as candidates for heart transplantation or LVAD for at least 6 months from randomization according to the opinion of the treating physician.
5. Women of childbearing potential (i.e., who have not undergone a hysterectomy or who have not been postmenopausal for at least 24 consecutive months) must commit either to abstain continuously from heterosexual sexual contact or to use at least one "highly effective" method of birth control (e.g., intrauterine device [IUD], hormonal contraception, tubal ligation, or partner's vasectomy) or two "effective" methods (e.g., latex condom, diaphragm, or cervical cap), beginning 4 weeks prior to screening and throughout study participation.

   Note: As alprostadil is not genotoxic and female sexual partners of male study participants are not likely to have substantial exposure via semen, there are no contraception requirements for men.
6. Patients must be willing and able to give written informed consent, including local data privacy consents, as required

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2026-10 (Estimated); Primary Completion 2029-11 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Time to all-cause mortality (defined as death, heart transplant, LVAD placement, mechanical circulatory support, or HF event(* hospitalization for HF or unplanned intravenous therapy for HF, ie diurectics, inotropes, vassopressors, or vasodilators.) | 6 months infusion
  To access the effect of continue 6-months ALP-1infusion at a fixed dose of at 500mcg/48 hr. in patinets with advanced heart failure with reduced ejection fraction(HrEF) compare to placebo.

SECONDARY OUTCOMES:
Secondary Efficacy and Safety Endpoints | 6 months
  . physcians review NYHA HF functional classification

CONTACTS AND LOCATIONS:
Overall Officials: Martin Huelsmann, MD, Principal Investigator — Medical university Vienna, Department of Cardiology; Noemi Pavo, MD PhD, Principal Investigator — Medical University Vienna, department of Cardiology
Locations (1):
- Medical university Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No